CLINICAL TRIAL: NCT01822782
Title: Abnormal Vaginal Flora and Vaginal Lesions at Delivery: is There a Relationship?
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2013/LB-01
Record Dates: First submitted 2013-03-28; First posted 2013-04-02 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2015-03

CONDITIONS: Vaginal Lesion
Keywords: Perineal tear; Perineal lesion; Vaginal flora; Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Cases: The study population consists of all consecutive women meeting inclusion/exclusion criteria and delivering at the Nîmes University Hospital, France during an inclusion period of 6 months. "Cases" are classified as those with a vaginal lesion due to delivery.
  Interventions: Biological: Bacteriological analysis of vaginal sample
- Controls: The study population consists of all consecutive women meeting inclusion/exclusion criteria and delivering at the Nîmes University Hospital, France during an inclusion period of 6 months. "Controls" are classified as those without a vaginal lesion due to delivery.
  Interventions: Biological: Bacteriological analysis of vaginal sample

INTERVENTIONS:
Biological: Bacteriological analysis of vaginal sample — Bacteriological analysis of vaginal sample

SUMMARY:
The main objective of this study is to assess whether the presence of abnormal vaginal flora (intermediate flora or vaginosis) is a risk factor for vaginal lesions at the time of delivery. For this, the primary endpoint will be the proportion of vaginal lesions according to the presence or absence of abnormal vaginal flora.

A more precise qualitative and quantitative study of vaginal flora isolated from pregnant women and its association with vaginal lesions will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a gestational age > 34 weeks delivering at the Nîmes University Hospital

Exclusion Criteria:

* Patient under judicial protection
* Adult patient under any kind of guardianship
* Patient refuses participation

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population consists of all consecutive women meeting inclusion/exclusion criteria and delivering at the Nîmes University Hospital, France during an inclusion period of 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Actual)
Dates: Start 2013-06; Primary Completion 2013-12-06 (Actual); Study Completion 2013-12-06 (Actual)

PRIMARY OUTCOMES:
Presence/absence of a vaginal lesion due to delivery | Upon delivery (Day 0)
Record of abnormal vaginal flora (presence/absence of Nugent's score > 3) in patient's medical file | Upon delivery (Day 0)
  Record of routine analysis of vaginal samples during pregnancy will be used.

SECONDARY OUTCOMES:
Recorded qualitative and quantitative analysis of vaginal flora in patient's file | Upon delivery (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie Becerra, Sage Femme, Principal Investigator — Centre Hospitalier Universitaire de Nîmes; Jean-Philippe Lavigne, MD, PhD, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, France

REFERENCES:
- [Result] Letouzey V, Bastide S, Ulrich D, Beccera L, Lomma M, de Tayrac R, Lavigne JP. Impact of Bacterial Vaginosis on Perineal Tears during Delivery: A Prospective Cohort Study. PLoS One. 2015 Nov 6;10(11):e0139334. doi: 10.1371/journal.pone.0139334. eCollection 2015. PMID 26544959